CLINICAL TRIAL: NCT06607913
Title: BCCMA: Recovery of Aged Muscle After Disuse Atrophy (REMEDY): Exercise and Monitoring With Post-Hospitalization Muscle Atrophy to Sustain Intrinsic Capacity and Strength (EMPHASIS)
Brief Title: Exercise and Monitoring With Post-Hospitalization Muscle Atrophy to Sustain Intrinsic Capacity and Strength
Acronym: EMPHASIS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CAMM-005-23F
Record Dates: First submitted 2024-09-19; First posted 2024-09-23 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Chronic Kidney Disease (CKD)
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Parallel study design features a Cohort Arm who will undergo regular assessments and observations for a minimum of 2 years. Participants who are hospitalized during the course of the study will undergo random assignment to an Exercise Group or a Usual Care group for 16-weeks.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Exercise (Experimental): The participants will exercise 2 days a week for 16 weeks. The exercises will include 4 movements: squats, shoulder press, seated row, and bicep curl focusing on internal load and contraction velocity.
  Interventions: Other: Exercise
- Usual Care (No Intervention): Participants will not have any study intervention visits for usual care.

INTERVENTIONS:
Other: Exercise — The participants will exercise 2 days a week for 16 weeks. The exercises will include 4 movements: squats, shoulder press, seated row, and bicep curl focusing on internal load and contraction velocity.
  Arms: Exercise

SUMMARY:
The aging Veteran population has more frequent inpatient hospitalization than non-Veterans. In addition, older Veterans have an inability to fully recover muscle mass and function after hospital-acquired weakness. The problem of hospital-acquired weakness is greatly increased in at-risk Veteran populations such as those with chronic kidney disease (CKD). The purpose of this collaborative study involving Denver and Baltimore VAMC sites is to improve health through the detection and rehabilitation management of hospital-acquired weakness in those with CKD. The study goals include identifying and monitoring the optimal muscle assessment sites in clinical settings, examining how muscle health impacts length of hospital stay and physical resilience, and determining how home-based and supervised exercise comparatively addresses post-hospitalization physical resilience using performance tests and Veteran feedback.

DETAILED DESCRIPTION:
This condition, known as disuse muscle atrophy, poses a substantial challenge to the health and well-being of individuals, particular those hospitalized. To tackle this problem , the project focuses on a specific group of individuals particularly vulnerable to this issues: Veterans with chronic kidney disease (CKD). This disease affects a substantial population of over 500,000 Veterans, leading to a progressive decline in mobility, unfavorable changes in lean body mass, and heightened hospitalization rates. To comprehensively address this concern, the project indents to develop and implement assessment and intervention strategies tailored to the target cohort's needs. By concentrating on Veterans with CKD, the project seeks to generate approaches that can be widely applied to address muscle atrophy among individuals with similar conditions. To achieve this, the project twill commence by establishing a baseline cohort of Veterans with Stage 3 and 4 CKD at two distinct Veterans Affairs sites located in Denver and Baltimore. Upon enrollment, the Veterans muscles health will be assessed, encompassing various dimensions such as strength, lean muscle mass, muscle composition, mobility, and intrinsic capacity. This comprehensive evaluation will provide a snapshot of their pre-hospitalization muscle health. Subsequently, the enrolled Veterans will be closely monitored for at least two years. The project's approach involves conducting regular assessments of their muscle health every six months. Additionally, the participating Veterans will provide information about their strength and functional status every quarter, facilitated through a smartphone application. A particular noteworthy aspect of the project is its inclusion of a pragmatic rehabilitation intervention trail. Veterans who experience hospitalization during the study will have the opportunity to participate in this trial. They will be assigned to either a supervised flywheel strengthening exercise group or receive usual care over 16 weeks. This intervention trial aims to assess the effective ness of targeted exercise in mitigating the effects of disuse muscle atrophy post-hospitalization. The overarching design of the project encompasses three main objectives:

Aim 1: Identify effective muscle assessment sites for disuse muscle atrophy. Aim 2: Assess if standardized intrinsic capacity and physical resilience assessments predict hospital outcomes. The investigators anticipate that physical resilience scores will improve hospitalization and strength outcomes predictions.

Aim 3: Evaluate a supervised flywheel exercise program against usual care. Both groups are expected to improve, with the supervised group have better results.

ELIGIBILITY:
Inclusion Criteria:

* Age > 55 years
* Diagnosis of stage 3-4 CKD or an eGFR of <45 mL/min/1.73m2

Exclusion Criteria:

* Cardiovascular risk: Poorly controlled hypertension (>160/100)

  * Coronary event in past 6 months
  * Class III or IV CHF
  * symptomatic angina at rest or during exercise
  * Syncope in past year, without known resolution of cause
* COPD requiring home oxygen
* Contraindications to resistance training, including history of intracranial or retinal bleeding; Diabetes with active proliferative retinopathy
* History of significant spinal osteoarthritis or spinal stenosis
* Dementia (on medical record review or mini-mental status exam score)

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2025-04-11 (Actual); Primary Completion 2028-09-30 (Estimated); Study Completion 2029-09-30 (Estimated)

PRIMARY OUTCOMES:
Vastus Lateralis Muscle Thickness | 4 month, 10 month
  A measure of the Vastus Lateralis muscle will be examined using ultrasound technology to determine the muscle size, quality, and composition. Post-intervention levels will be compared to 6 months after the cessation of the intervention.
Function | 4 month, 10 month
  The short physical performance battery test is a function measure that utilizes 3 tasks scores 0-4 (total possible score of 12) to determine functional status and lower extremity function. Pre-test scores will be compared to post intervention test scores.
Lower Extremity Strength - Isometric Strength | 4 month, 10 month
  A measures of maximal isometric muscle strength produced in knee extensor muscles will be assessed with a Biodex device. Post-intervention levels will be compared to 6 months after the cessation of exercise.
Upper Extremity Strength - Grip Strength | 4 month, 10 month
  A measures of maximal isometric muscle strength produced in upper extremity muscles will be assessed by grip strength. Post-intervention levels will be compared to 6 months after the cessation of exercise.

SECONDARY OUTCOMES:
Rectus Femoris Muscle Thickness | 4 month, 10 month
  A measure of the Rectus Femoris muscle will be examined using ultrasound technology to determine the muscle size, quality, and composition. Post-intervention levels will be compared to 6 months after the cessation of the intervention.
Bicep Brachii Muscle Thickness | 4 month, 10 month
  A measure of the Bicep Brachii muscle will be examined using ultrasound technology to determine the muscle size, quality, and composition. Post-intervention levels will be compared to 6 months after the cessation of the intervention.
Middle Deltoid Muscle Thickness | 4 month, 10 month
  A measure of the Middle Deltoid muscle will be examined using ultrasound technology to determine the muscle size, quality, and composition. Post-intervention levels will be compared to 6 months after the cessation of the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Harris-Love, DSc MPT BS, Principal Investigator — Rocky Mountain Regional VA Medical Center, Aurora, CO
Locations (2):
- United States (2):
  - Rocky Mountain Regional VA Medical Center, Aurora, CO, Aurora, Colorado
  - Baltimore VA Medical Center VA Maryland Health Care System, Baltimore, MD, Baltimore, Maryland

IPD SHARING:
Plan to Share IPD: No